CLINICAL TRIAL: NCT02276326
Title: Title Effect of Microbial Translocation and Supplementation With the Probiotic VSL#3 on Neuro-cognitive Functions of HIV Positive Patients Receiving HAART
Brief Title: Effects of VSL#3 on Neuro-cognitive Profile of HIV Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Gabriella D'Ettorre, PhD, Azienda Policlinico Umberto I
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VSL-Dett 2014
Record Dates: First submitted 2014-10-17; First posted 2014-10-28 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: HIV Seropositivity; ART
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VSL#3 sachets (Experimental): VSL#3 is a mix of lactic acid bacteria and bifidobacteria (original De Simone's formulation)
  Interventions: Dietary Supplement: VSL#3 sachets

INTERVENTIONS:
Dietary Supplement: VSL#3 sachets — 4 sachets a day for 4 months

SUMMARY:
Aim of the study is to evaluate the effects of a change in the intestinal microflora on the neuro-cognitive profile of patients with HIV infection receiving HAART treatment. Improvements will be evaluated with questionnaires on Quality of life and Cognitive and Behavior function.

20 patients will be enrolled and will receive 4 sachets of VSL#3 per day.

DETAILED DESCRIPTION:
The HIV virus has a marked tropism for the central nervous system. In 1986, the term AIDS Dementia Complex (ADC) has been coined which includes in a single syndrome, a whole series of severe neurologic manifestations, characterized by cognitive, motor and behavioral disorders.

The introduction of HAART has led to a profound change of the neurological HIV-mediated profile.

The increased morbidity that occurs in HIV patients on antiretroviral therapy is related to inflammatory processes and cardiovascular diseases, resulting from the damage of the mucosa of the gastrointestinal tract.

The massive depletion of CD4 T cells in the GI tract, low frequencies of CD4 and CD8 T producing IL-17, apoptosis of enterocytes (resulting in structural damage to the barrier of the GI tract) and the increase in intestinal permeability, are all manifestations of progressive HIV infection in humans.

The main consequence of the structural and functional disruption of the enteric mucosal barrier is constituted by the passage into the systemic circulation of products of microbial origin including the lipopolysaccharide (LPS), a phenomenon known as "microbial translocation" (MT). A direct consequence of MT is the increase in the levels of systemic innate and adaptive immune activation. The alteration of the intestinal mucosa also involves changes in the composition of the local microbial flora, event that changes the normal balance of the so-called axis "brain-gut", the function of this axis is in fact influenced by metabolic products of the resident bacterial flora.

The disturbance of this balance can cause diseases such as anxiety and depression

It's scientifically proved the importance that the intestinal microflora (in particular bifidobacteria and lactobacilli) plays in relation to the multiple tasks that you can perform, such as:

1. reduction of the intraluminal pH by the production of lactic acid, acetic acid and other organic acids;
2. production of nutrients (short chain fatty acids, arginine, glutathione, vitamins, etc..) of extreme importance for the normal trophism of the intestinal mucosa;
3. stimulation of the immune system and in particular: the macrophage activity, cytokine production, natural killer activity, the proliferation of lymphocytes, the production of IgA;
4. competition with pathogens for nutrients and adhesion in the gut epithelium;
5. production of bacteriocins;
6. modulation of the inflammatory response.

The intestinal microflora, therefore, plays a metabolic activity of enormous importance both on a purely nutritional level and for the maintenance of an efficient barrier activity of the intestinal mucosa, which together with the modulation of local and systemic immune response, is fundamental for the protection of the host organism.

VSL # 3 (original De Simone's formulation) is a probiotic preparation at a high concentration (450 billion bacteria per sachet) consisting of: 4 strains of lactobacilli (L. acidophilus, L. paracasei, L. delbrueckii subs. bulgaricus, L. plantarum), 3 strains of bifidobacteria: (B. breve, B. infantis, B. longum) and one strain of Streptococcus thermophilus. This product is able to colonize the intestine and to modulate the intestinal microflora. The efficacy of VSL#3 was proven in the treatment of inflammatory bowel diseases (ulcerative colitis, pouchitis mainly) as well as in the prevention or treatment of various gastrointestinal disorders such as diarrhea from rotavirus, traveler's diarrhea, diarrhea after antibiotic therapy and radiotherapy. Several studies have demonstrated the efficacy of VSL# in chronic diseases of the liver (steatosis, steatohepatitis, NAFLD, etc ...). Recently Klatt et al demonstrated that treatment antiretroviral (ARV) in association with VSL#3 at a dose of 225 billion / day) and prebiotics (inulin), for a period of 5 months in a population of macaques resulted in an increased reconstruction and functionality of CD4 + cells and a reduced fibrosis at the level of lymphoid follicles of the colon mucosa, compared to the group of macaques treated with ARV therapy alone. A decrease of immuno-activation of CD4 + cells in the mucosa of the colon and a decrease of plasma levels of D-dimers was observed in macaques treated with ARV therapy in combination with probiotic + prebiotic, compared to the group control. It is good to emphasize that the dimers are biomarkers of inflammation-related cardiovascular disease in HIV patients treated with ARV therapy (Klatt, 2013). All this clearly leads to an improvement of the immunity of the gastrointestinal tract, with consequent reduction of inflammatory processes and improving the prognosis of HIV infection.

SUB-STUDIES:

Given the implication of chronic immune activation and intestinal microbiota alterations in HIV-1 disease progression and non-AIDS related damages, we considered that supplementing antiretroviral therapy in HIV-1 infected patients with a probiotic mixture might promote beneficial effects in the restoration of HIV related damage of the intestinal epithelium and Gut-Associated Lymphoid Tissue (GALT).

To explore the potential impact of probiotics on intestinal damage, we have designed a substudy that analyzes the following parameters: T cell activation and CD4+ and CD8+ T-cell subsets expressing interferon (IFN)γ (Th1, Tc1) or interleukin (IL)-17A (Th17, Tc17) by multi-parameter flow cytoflorimetric analysis, histological and immunohistochemical analysis of intestinal biopsies TUNEL assay to determine enterocytes apoptosis index.

Addendum: - Amendment 1 (enrollment of naive patients) Amendment 2 (enrollment of healty controls) Amendment 3 (enrollment of control group) Amendment 4 (supplementation for 6 months)

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years of age
* In HAART with HIV RNA <50cp/mL, with CD4 counts> 400 cells / mm
* Availability to release informed consent

Exclusion Criteria:

* Patients with known allergy or intolerance to VSL#3
* Chronic inflammatory bowel diseases
* Drug addiction
* Use of antibiotics or probiotics during the 3 weeks prior the enrollment
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Delta of scores of questionnaires on quality of life | 4 months
  HIV dementia-scale, Beck Depression Inventory BDI-II, State Trait Anxiety Inventory (STAI Y 1 - Y2), the questionnaire for the assessment of quality of life in persons with HIV infection (ISS-QoL)
Delta of scores of questionnaires on cognitive functions | 4 months
  HIV dementia-scale, Beck Depression Inventory BDI-II, State Trait Anxiety Inventory (STAI Y 1 - Y2), the questionnaire for the assessment of quality of life in persons with HIV infection (ISS-QoL)
Delta of scores of questionnaires on behavioral functions | 4 months
  HIV dementia-scale, Beck Depression Inventory BDI-II, State Trait Anxiety Inventory (STAI Y 1 - Y2), the questionnaire for the assessment of quality of life in persons with HIV infection (ISS-QoL)

SECONDARY OUTCOMES:
Delta of value of serum lipopolysaccharide (LPS) | between time 0 and after 4 months of assumption of VSL#3

OTHER OUTCOMES:
Delta of Cluster of Differentiation 14 (CD14)+ in blood (T0-T1) | between time 0 and after 4 months of assumption
Delta of value of serum lipopolysaccharide binding protein (LBP) | between time 0 and after 4 months of assumption
Delta of value of serum EndoCAb | between time 0 and after 4 months of assumption
Delta of value of serum hs-CRP | between time 0 and after 4 months of assumption
Delta of value of serum IL-6 | between time 0 and after 4 months of assumption
Delta of value of serum TNFa | between time 0 and after 4 months of assumption
Delta of value of serum MIP-lb | between time 0 and after 4 months of assumption

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella D'Ettorre, Principal Investigator — Policlinico Umberto I Hospital
Locations (1):
- Policlinico Umberto I Hospital, Rome, Italy

REFERENCES:
- [Result] Ceccarelli G, Brenchley JM, Cavallari EN, Scheri GC, Fratino M, Pinacchio C, Schietroma I, Fard SN, Scagnolari C, Mezzaroma I, Vullo V, d'Ettorre G. Impact of High-Dose Multi-Strain Probiotic Supplementation on Neurocognitive Performance and Central Nervous System Immune Activation of HIV-1 Infected Individuals. Nutrients. 2017 Nov 21;9(11):1269. doi: 10.3390/nu9111269. PMID 29160817
- [Result] Ceccarelli G, Fratino M, Selvaggi C, Giustini N, Serafino S, Schietroma I, Corano Scheri G, Pavone P, Passavanti G, Alunni Fegatelli D, Mezzaroma I, Antonelli G, Vullo V, Scagnolari C, d'Ettorre G. A pilot study on the effects of probiotic supplementation on neuropsychological performance and microRNA-29a-c levels in antiretroviral-treated HIV-1-infected patients. Brain Behav. 2017 Jul 16;7(8):e00756. doi: 10.1002/brb3.756. eCollection 2017 Aug. PMID 28828217
- [Derived] Santinelli L, Ceccarelli G, Borrazzo C, Innocenti GP, Frasca F, Cavallari EN, Celani L, Nonne C, Mastroianni CM, d'Ettorre G. Sex-related differences in markers of immune activation in virologically suppressed HIV-infected patients. Biol Sex Differ. 2020 May 1;11(1):23. doi: 10.1186/s13293-020-00302-x. PMID 32357901